CLINICAL TRIAL: NCT01918904
Title: A Pilot Study to Evaluate Topical Sodium Thiosulfate Therapy for Calcinosis Cutis (STS-CALC)
Brief Title: A Pilot Study to Evaluate Topical Sodium Thiosulfate Therapy for Calcinosis Cutis
Acronym: STS-CALC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided not to proceed with this project. No participants were enrolled.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elaine Adams, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 205683
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Calcinosis Cutis
Keywords: calcinosis; sodium thiosulfate; topical treatment; connective tissue disease
MeSH Terms: conditions — Calcinosis Cutis; Calcinosis; Connective Tissue Diseases | interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Thiosulfate (Experimental): A small amount of 25% topical sodium thiosulfate cream twice daily (bid)
  Interventions: Drug: Sodium thiosulfate
- Placebo (Placebo Comparator): A small amount of topical zinc oxide and aquaphor cream twice daily (bid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium thiosulfate — A small amount of 25% topical sodium thiosulfate cream twice daily (bid)
  Arms: Sodium Thiosulfate
Drug: Placebo — A small amount of topical zinc oxide and aquaphor cream twice daily (bid)
  Arms: Placebo

SUMMARY:
Calcinosis cutis refers to a group of disorders characterized by calcium deposition in the skin (1). The disorders are classified according to etiology into the following types: dystrophic, metastatic, iatrogenic, and idiopathic (1,2). Dystrophic calcification occurs in the setting of varicosities, infection, tumors, and connective tissue disorders (1). The connective tissue disorders most commonly associated with calcinosis cutis are systemic sclerosis and dermatomyositis, although it has also been reported in patients with systemic lupus erythematosus, undifferentiated connective tissue disorder, and mixed connective tissue disorder (2). The pathophysiology of calcinosis cutis is not well understood, and there is a broad range of severity seen, from benign localized, small nodules to large, severely debilitating lesions (2). Although many therapies have been investigated for treatment of calcinosis cutis, including calcium channel blockers, colchicine, minocycline, intravenous immunoglobulin, and bisphosphonates, results have been mixed at best (2). Surgical removal is sometimes feasible in the case of a localized lesion, however, recurrence after surgery is common (2).

Recently, several authors have reported cases of dramatic resolution of dystrophic calcinosis cutis lesions with topical sodium thiosulfate preparations (1,3,4). Systemic sodium thiosulfate therapy is commonly used to treat calciphylaxis in patients with renal disorders with very few adverse events (1). A search of the literature to date yields no formal studies that aim to determine whether topical sodium thiosulfate is truly an effective therapy for calcinosis cutis. As a result, patients are often treated with therapies that are unproven or ineffective and their calcinosis cutis eventually leads to significant pain and disability.

Research Question:

Does treatment of dystrophic calcinosis cutis with topical sodium thiosulfate result in diminution of the lesion and associated pain?

Objective:

The objective of this pilot study is to investigate whether topical sodium thiosulfate is an effective therapy for calcinosis cutis. This study will also determine the feasibility of our protocol and provide information to help direct a future full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen by the Division of Rheumatology at Loyola Outpatient Center in Maywood, Illinois (IL), Oak Brook Terrace Outpatient Center in Oakbrook, IL, and Burr Ridge Outpatient Center in Burr Ridge, IL.
* Male and female patients 18 years old and above
* Patients with at least 2 distinct calcinosis cutis lesions separated by at least 10 inches, that are a minimum of 2 millimeters (mm) in diameter, and identifiable on physical exam and ultrasound, such that one lesion may be used as an internal control lesion
* Patients on calcium channel blockers, bisphosphonates, prednisone, and colchicine will be included

Exclusion Criteria:

* Patients with calcinosis cutis lesions that appear actively infected (i.e., exhibiting purulent drainage and malodor) will not be included
* Patient with concomitant use of systemic intravenous sodium thiosulfate for treatment of calciphylaxis will not be included
* Patients with hypercalcemia will not be included
* Patients who are pregnant or breastfeeding will not be included
* Patients who are allergic to sulfa and/or zinc will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in calcinosis cutis lesion size from week 0 to week 12 for the experimental arm versus placebo arm | After 12 weeks of treatment
  Definition: Calcinosis cutis lesion. Change Calculation Details: The lesion size will be evaluated at week 0 and again at week 12. Continuous measurement of the lesion in millimeters (mm), where a decrease in diameter indicates improvement.

SECONDARY OUTCOMES:
Change in pain from week 0 to week 12 for the experimental arm versus placebo arm | After 12 weeks of treatment
  (1) Full Scale Name: 100mm Visual Analog Pain Scale (VAS). (2) Definition: The VAS is a pain scale. (3) Construct measured: Pain. (4) VAS Score Range: Raw scores may range from 0 to 10, where higher scores indicate worsening pain. (5) Change Calculation Details: Ordinal measure comparing pain from Baseline (week 0) to Week 12 for the experimental versus placebo arm
Change in pain from week 0 to week 24 for the experimental arm versus placebo arm | After 24 weeks of treatment
  (1) Full Scale Name: 100mm Visual Analog Pain Scale (VAS). (2) Definition: The VAS is a pain scale. (3) Construct measured: Pain. (4) VAS Score Range: Raw scores may range from 0 to 10, where higher scores indicate worsening pain. (5) Change Calculation Details: Ordinal measure comparing pain from Baseline (week 0) to Week 24 for the experimental versus placebo arm
Change in calcinosis cutis lesion size from week 0 to week 24 for the experimental arm versus placebo arm | After 24 weeks of treatment
  Definition: Calcinosis cutis lesion. Change Calculation Details: The lesion size will be evaluated at week 0 and again at week 24. Continuous measurement of the lesion in millimeters (mm), where a decrease in diameter indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Adams, M.D., Principal Investigator — Loyola University; Melissa R Bussey, M.D., Study Director — Loyola University

REFERENCES:
- [Background] Bair B, Fivenson D. A novel treatment for ulcerative calcinosis cutis. J Drugs Dermatol. 2011 Sep;10(9):1042-4. PMID 22052275
- [Background] Gutierrez A Jr, Wetter DA. Calcinosis cutis in autoimmune connective tissue diseases. Dermatol Ther. 2012 Mar-Apr;25(2):195-206. doi: 10.1111/j.1529-8019.2012.01492.x. PMID 22741938
- [Background] Ratsimbazafy V, Bahans C, Guigonis V. Dramatic diminution of a large calcification treated with topical sodium thiosulfate. Arthritis Rheum. 2012 Nov;64(11):3826. doi: 10.1002/art.34628. No abstract available. PMID 22806424
- [Background] Wolf EK, Smidt AC, Laumann AE. Topical sodium thiosulfate therapy for leg ulcers with dystrophic calcification. Arch Dermatol. 2008 Dec;144(12):1560-2. doi: 10.1001/archderm.144.12.1560. No abstract available. PMID 19075137